CLINICAL TRIAL: NCT04820270
Title: Infusion of Autologous T Regulatory Cells (T Reg) at the Time of Transplantation of Allogenic Islets of Langerhans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Nordic Network For Clinical Islet Transplantation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AutoTregIsl
Record Dates: First submitted 2021-03-16; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Type1diabetes
Keywords: Transplantation; Islets of Langerhans; T regulatory Cells (autologous)

STUDY DESIGN:
Intervention Model Description: Single arm feasibility and safety study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Tregs in allogenic islet transplantation (Experimental): Autologous Tregs are given simultaneously to the patient with the islets
  Interventions: Other: Autologous T regulatory cells

INTERVENTIONS:
Other: Autologous T regulatory cells — Enriched autologous T regulatory cells are given back to the patient at the time of islet transplantation

SUMMARY:
Open single armed study to investigate safety and feasibility of administrating autologous T regulatory cells at the time of allogenic islet transplantation.

DETAILED DESCRIPTION:
Open single armed study to investigate safety and feasibility of administrating autologous T regulatory cells at the time of allogenic islet transplantation. Patients are recruited from the waiting list for islet transplantation within The Nordic Network for Clinical Islet Transplantation. Patients included in the study will undergo apheresis while on the waiting list. T regulatory cells will be sorted out and frozen. Autologous, non modified T regs will then be infused simultaneously intraportally with the islet graft at transplantation. Patients will be followed for safety and efficacy regarding the islet transplantation over three months

ELIGIBILITY:
Inclusion Criteria:

* Patient must be registered on the waiting list within The Nordic Network for Clinical Islet Transplantation
* Type 1 diabetes with diagnosed <40years of age and with>5 years of exogenous insulin use
* C peptide < 0.1 nmol/L at MMTT if no previous islet transplant
* Adequate previous treatment by an experienced diabetologist
* Patient must understand and be able to sign an informed consent

Exclusion Criteria:

* Patient with a previous transplant other than islets
* Patient with an BMI>30
* Patient with an need of more than 1U/kg of insulin per 24h
* Repeated abnormal liver function tests
* non stable retinopathy
* known abnormalities in coagulation
* known malignancies
* non stable heart conditions
* active infections
* serological proof of hepatitis B or C or HIV
* signs of portal hypertension
* patients that are pregnant, breast feeding or aim to become pregnant during the study period
* patients with a PRA > 20%, positive cross match or known DSA
* patients with conditions that the investigator would consider unsafe to combine with islet transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding | 0-1 days post transplant
  Number of patients with >20g/L reduction of haemoglobine and signs of bleeding shown by ultrasound post operative day 1
Thrombosis | 0-75 days post transplant
  Number of patients with thrombosis in portal veins shown by ultrasound post operative day 1 or later
Liver function | 0-75days
  Number of patients with an elevation of transaminases > 5 times upper normal level during follow up
Infections | 0-90 days post transplantation
  Number of treatment requiering infections in each patient during follow up
Islet graft failure | day 75
  Number of patients with islet graft failure shown as C peptide <0.1 nmol/L fasting or <0.3 nmol/L (90min) at a MMTT day 75 or lack of improvement compared to baseline if transplanted before.
Immunization | 90 days post transplantation
  Number of patients with new anti HLA antibodies found at 90 days post transplantation compared to baseline

SECONDARY OUTCOMES:
Islet function | day 75
  Fraction of patients with a C-peptide level above 0.1 nmol/L fasting or 0.3 nmol/L (90min) at a MMTT day 75
Insulin independence | day 75
  Fraction of patients without need of exogeous insulin (ADA criteria) at day 75 post transplantation
HbA1c | day 75
  Mean reduction of HbA1c at day 75 compared to baseline(%)
Hypoglycemic unawareness | day 75
  Number of patients with a reduced Clarke hypoglycemia awareness score day 75 (+/-5) post transplantation compared to baseline
HbA1c and hypoglycemic unawareness combined | day 75
  Number of patients with both a HbA1c ≤ 6.5% (DCCT) and lack of severe hypoglycemia at day 75 post transplantation
PRA level | day 90
  Number of patients with a rise in PRA (panel reactive antibodies) with more than 10% at 90 days post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lundgren, MD, Principal Investigator — Karolinska University Hospital
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala